CLINICAL TRIAL: NCT05988008
Title: A Phase I Clinical Study of CCX168 in Japanese and Caucasian Healthy Adult Males
Brief Title: A Study of CCX168 in Japanese and Caucasian Healthy Adult Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CCX1101
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Anti-neutrophil Cytoplasmic Antibody-associated Vasculitis
Keywords: Human C5a receptor (C5aR); Vasculitis; Complement; Vascular disease
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Vasculitis; Vascular Diseases | interventions — avacopan

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A: Single Oral Dosing of CCX168 in Japanese Adult Males (Experimental): Healthy Japanese adult males will receive 1 of 3 single oral doses of CCX168 (10 mg, 30 mg or 100 mg) or placebo. Each dose level will be administered under fasted conditions. Single doses of CCX168 30 mg will be administered under fasted and fed conditions.
  Interventions: Drug: CCX168; Drug: Placebo
- Cohort B: Multiple Oral Dosing of CCX168 in Japanese Adult Males (Experimental): Healthy Japanese adult males will receive 1 of 2 oral doses of CCX168 (30 mg or 50 mg) or placebo twice-daily for 7 days under fed conditions.
  Interventions: Drug: CCX168; Drug: Placebo
- Cohort C: Single Oral Dosing of CCX168 in Caucasian Adult Males (Experimental): Healthy Caucasian adult males will receive 1 of 2 single oral doses of CCX168 (10 mg or 30 mg) or placebo under fasted conditions.
  Interventions: Drug: CCX168; Drug: Placebo
- Cohort D: Multiple Oral Dosing of CCX168 in Caucasian Adult Males (Experimental): Healthy Caucasian adult males will receive an oral dose of CCX168 30 mg or placebo twice-daily for 7 days under fed conditions.
  Interventions: Drug: CCX168; Drug: Placebo

INTERVENTIONS:
Drug: CCX168 — Administered orally.
  Other Names: Avacopan
Drug: Placebo — Administered orally.

SUMMARY:
The objectives of the study will be to investigate the safety and pharmacokinetics of a single oral administration and a twice-daily multiple oral administration of CCX168 in Japanese healthy adult males; and to compare the pharmacokinetics of a single oral administration and a twice-daily multiple oral administration of CCX168 between Japanese and Caucasian healthy adult males.

ELIGIBILITY:
Inclusion Criteria:

* Japanese and Caucasian healthy males aged 20 to 45 years inclusive (at the time of obtaining informed consent);
* Body Mass Index (body weight [kg]/squared height [m^2]): 18.5 kg/m^2 or more and less than 25 kg/m^2 for Japanese males or between 18.5 and 29 kg/m^2 for Caucasian males (at the time of screening visit);
* Body weight: 50 kg or more and less than 90 kg (at the time of screening visit).

Exclusion Criteria:

* Participants with any abnormal findings (e.g., clinical laboratory test values outside the reference range) during the physical examination and other tests (vital signs, 12-lead ECG and clinical laboratory tests) that are judged by the principal investigator or subinvestigator to be clinically significant;
* Participants who test positive for immunological tests (hepatitis B surface antigen, hepatitis C virus antibody, serological reaction of syphilis, and human immunodeficiency virus antigen and antibody);
* Participants with a history of drug allergy;
* Participants who are a habitual alcohol drinker with an average pure alcohol intake of over 40 g/day;
* Participants who test positive for abuse of phencyclidines, benzodiazepines, cocaine, stimulants, cannabis, morphine, barbiturates, and tricyclic antidepressants during urine drug testing;
* Male participant who do not agree to use adequate contraception for a period from a start of the investigational product administration to 12 weeks after the final administration of the investigational product;
* Participants with a QTcF intervals of 450 msec or greater in the 12-lead ECG at the time of the screening visit and/or Day -1;
* Participants who consumed tobacco or a nicotine patch/gum within 12 weeks prior to the investigational product administration;
* Participants who received other prescription medications or over-the-counter medications (including vitamins and energy drinks) within 2 weeks prior to the investigational product administration (excluding topical formulation that is not expected systemic action);
* Participants who received any supplements (Saint John's wort [Hypericum perforatum] etc.) that have been reported to affect the pharmacokinetics of concomitant use of drugs within 2 weeks prior to the investigational product administration;
* Participants who received a grapefruit and an orange that contain the component inhibiting CYP3A4 or the food and drink containing these fruits within 1 week prior to the investigational product administration;
* Participants who received other investigational products within 16 weeks prior to the investigational product administration;
* Participants who donated more than 200 mL of blood (donation of whole blood, plasma components or platelets, etc.) within 4 weeks or more than 400 mL within 16 weeks prior to the investigational product administration;
* Participants who performed excessive exercise with symptoms of fatigue or muscle pain within 1 week prior to the investigational product administration;
* Participants who are judged by the principal investigator or subinvestigator as inappropriate for inclusion in this study.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events | Up to 14 days
Number of Participants Experiencing Adverse Drug Reactions | Up to 14 days
Number of Participants Experiencing Clinically Significant Changes in Vital Sign Parameters | Up to 14 days
Number of Participants Experiencing Clinically Significant Changes in Electrocardiogram (ECG) Parameters | Up to 14 days
Number of Participants Experiencing Clinically Significant Changes in Clinical Laboratory Parameters | Up to 14 days
Maximum Plasma Concentration (Cmax) of CCX168 | Up to 14 days
Cmax of CCX168-M1 (Metabolite) | Up to 14 days
Time of Cmax (tmax) of CCX168 | Up to 14 days
Tmax of CCX168-M1 | Up to 14 days
Area Under the Plasma Concentration Time Curve (AUC) from Time 0 to Infinity (AUC0-inf) of CCX168 | Up to 14 days
AUC0-inf of CCX168-M1 | Up to 14 days
AUC from Time 0 to Time of Last Measurable Plasma Concentration (AUC0-tz) of CCX168 | Up to 14 days
AUC0-tz of CCX168-M1 | Up to 14 days
AUC During a Dosing Interval of CCX168 | Cohorts B and D only: Up to Hour 12 post-dose on Days 1 - 7
AUC During a Dosing Interval of CCX168-M1 | Cohorts B and D only: Up to Hour 12 post-dose on Days 1 - 7
Terminal Elimination Half-life of CCX168 | Up to 14 days
Terminal Elimination Half-life of CCX168-M1 | Up to 14 days
Apparent Oral Clearance of CCX168 | Up to 14 days
Apparent Volume of Distribution During the Terminal Phase of CCX168 | Up to 14 days
Mean Residence Time to Infinity of CCX168 | Up to 14 days
Accumulation Ratio of CCX168 | Cohorts B and D only: Up to 14 days
Accumulation Ratio of CCX168-M1 | Cohorts B and D only: Up to 14 days
Trough Plasma Concentration at the End of Dosing Interval of CCX168 | Cohorts B and D only: Up to 14 days
Trough Plasma Concentration at the End of Dosing Interval of CCX168-M1 | Cohorts B and D only: Up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Sumida Hospital, SOUSEIKAI Global Clinical Research Center, Sumida City, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com